CLINICAL TRIAL: NCT03653598
Title: BLITZ Atrial Fibrillation
Acronym: BLITZ-AF
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K16
Record Dates: First submitted 2018-08-09; First posted 2018-08-31 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AF patients: Patients with Atrial Fibrillation
  Interventions: Other: Atrial Fibrillation

INTERVENTIONS:
Other: Atrial Fibrillation — Data collection on Atrial Fibrillation

SUMMARY:
Management strategies for AF have made many advances over the last decade but there is still a great heterogeneity in the management of AF and it remains unclear how often clinicians adhere to current guidelines.

A survey of an updated AF management would enable a timely assessment of implementation of current International guidelines, allow monitoring of early management of AF when a patients is admitted in a Emergency Room (ER) and Cardiology Unit.

DETAILED DESCRIPTION:
Multicentre, observational study. 200 Italian Hospitals fully representing the Italian cardiology reality in terms of geographical distribution and level of hospital technology.

Data collection in ER: Data on AF and Atrial Flutter episodes in ER will be collected retrospectively by checking the records of ER without collection of any data that can allow to identify the patients. These data will be collected under the responsibility of the Cardiology Departments consecutively for 4 weeks.

Data collected in Cardiology: these data will be collected under the responsibility of the Cardiology Departments for 12 weeks consecutively.

ELIGIBILITY:
Inclusion Criteria:

* All patients with AF, admitted to cardiology wards for an urgent or planned hospitalization.
* All patients admitted in a Day Hospital regimen for treatment of AF The diagnosis of AF must be confirmed by ECG.
* Signed Patient Inform Consent.

Exclusion Criteria:

* The qualifying episode of AF was not documented with an ECG.
* Age <18 years.
* Patients with AF as a complication of an acute coronary syndrome (within 1 week from symptoms onset).
* Patients with AF associated with cardiothoracic surgery (within 1 week from surgery).
* Concomitant participation in other studies that can modify the diagnostic and/or therapeutic treatments.
* Patients already enrolled in BLITZ-AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive hospitalized patients with Atrial Fibrillation
Sampling Method: Probability Sample
Enrollment: 4125 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of admissions of patients with AF | Enrollemnt
  Number of admissions to the ER and cardiology wards of patients with AF
Rate or rhythm control strategy | Baselane study completion - average 1 week
  Percentage of patients in rate or thythm control therapy
Antithrombotic strategies | Baselane study completion - average 1 week
  Rate of use of oral antithrombotic strategies

SECONDARY OUTCOMES:
Admission to the ER for atrial flutter | Enrollment
  Number of admission to the ER for atrial flutter
Patients regularly followed up by the cardiology centers | 12 months
  Rate of patients regularly followed up by the cardiology centers
Adherence to the 1A recommendations of current guidelines | 12 months
  Rate of adherence to the 1A recommendations of current guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gulizia, MD, Study Chair — Heart Care Foundation
Locations (154):
- Italy (154):
  - Ospedale San Giovanni Di Dio - Uo Cardiologia E Utic, Agrigento, AG
  - Ospedale Santo Spirito - Sc Cardiologia, Casale Monferrato, AL
  - Ospedale Civile Profili - U.O. Cardiologia, Fabriano, AN
  - Ospedale Di Jesi Carlo Urbani - U.O. Di Cardiologia, Iesi, AN
  - Ospedale Principe Di Piemonte - Uoc Cardiologia Utic, Senigallia, AN
  - Ospedale Generale Regionale-Po U. Parini - U.O. Cardiologia E Cure Intensive Card., Aosta, AO
  - Ospedale Gen.Le Prov.Le C.G. Mazzoni - Sc Cardiologia, Ascoli Piceno, AP
  - Ospedale Valdichiana Santa Margherita - Uos Cardiologia E Hdu, Cortona, AR
  - Po Sant'Ottone Frangipane - U.O.C. Cardiologia - Utic, Ariano Irpino, AV
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Della Murgia - Fabio Perinei - S.C. Cardiologia-Utic, Altamura, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Policlinico - U.O. Di Cardiologia Ospedaliera, Bari, BA
  - Ospedale Umberto I - Uosd Di Cardiologia, Corato, BA
  - P.O. Don Tonino Bello - Uosd Cardiologia, Molfetta, BA
  - Iob - Policlinico San Marco - U.O. Cardiologia, Osio Sotto, BG
  - Ospedale Civile - Sc Cardiologia, Belluno, BL
  - Ospedale Santa Maria Del Prato - U.O. Di Cardiologia, Feltre, BL
  - Azienda Ospedaliera G. Rummo - Cardiologia Interventistica E Utic, Benevento, BN
  - Ospedale Maggiore - Uo Di Cardiologia, Bologna, BO
  - Ospedale Bellaria - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Ospedale Civile Dario Camberlingo - U.O. Di Cardiologia - Utic, Francavilla Fontana, BR
  - Ospedale Di Gardone Val Trompia - Ssvd Cardiologia, Gardone Val Trompia, BS
  - Osp. Andria Canosa - Po Andria - Cardiologia - Utic, Andria, BT
  - Ospedale Monsignor Angelo R. Di Miccoli - Unita' Operativa Di Cardiologia, Barletta, BT
  - Ospedale Vittorio Emanuele Ii - Cardiologia, Bisceglie, BT
  - Ospedale Generale Regionale - Divisione Di Cardiologia, Bolzano, BZ
  - Presidio Ospedaliero Ss Trinita' - Sc Di Cardiologia, Cagliari, CA
  - Az. Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia-Utic, Caserta, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Presidio Ospedaliero San Rocco - U.O.C. Cardiologia - Utic, Sessa Aurunca, CE
  - Ospedale 'Renzetti' - Cardiologia E Utic, Lanciano, CH
  - Ospedale S. Elia - U.O.C Cardiologia - Utic, Caltanissetta, CL
  - Ospedale Moriggia Pelascini - Unita' Operativa Di Cardiologia, Gravedona, CO
  - Ospedale Maggiore - U.O. Cardiologia E Utic, Crema, CR
  - Ospedale Di Cremona - Uo Di Cardiologia, Cremona, CR
  - Ospedale Spoke Paola- Cetraro Po Paola - Utic Cardiologia, Paola, CS
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania, CT
  - Azienda Ospedaliera Cannizzaro -, Catania, CT
  - Ospedale G. Basilotta - U.O.C. Di Cardiologia, Nicosia, EN
  - Ospedale Ss. Annunziata - U.O. Di Cardiologia, Cento, FE
  - Ospedale Civile Giuseppe Tatarella - U.O. Di Cardiologia - Utic, Cerignola, FG
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale Civile Augusto Murri - U.O. Cardiologia, Fermo, FM
  - Ospedale Civile San Polo - S.O.C. Cardiologia, Monfalcone, GO
  - Ospedale San Leopoldo Mandic - Cardiologia - Ucc, Merate, LC
  - Presidio Ospedaliero F. Ferrari - Cardiologia - Utic, Casarano, LE
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia-Utic, Copertino, LE
  - Ospedale Santa Caterina Novella - U.O. Di Cardiologia, Galatina, LE
  - Ospedale Civile Sacro Cuore Di Gesu' - Uo Cardiologia Utic, Gallipoli, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic, Scorrano, LE
  - Ospedale Villamarina - Cardiologia E Utic, Piombino, LI
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale Carate Brianza - Cardiologia- Carate Brianza/Giussano, Carate Brianza, MB
  - Ospedale San Gerardo - U.O. Cardiologia-Utic, Monza, MB
  - Policlinico Di Monza - Uo Cardiol. Clinica E Scompenso Cardiaco, Monza, MB
  - Presidio Osp. Di Civitanova Marche - Sc Cardiologia, Civitanova Marche, MC
  - Ospedale Barone Romeo - Divisione Di Cardiologia E Utic, Patti, ME
  - P.O. Sant'Agata Di Militello - Uoc Cardiologia, Sant'Agata di Militello, ME
  - Centro Cardiologico Monzino - Scompenso,Cardiologia Clinica, Riabilit., Milan, MI
  - Ospedale San Luca - Istituto Auxologico - U.O. Cardiologia, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia-Ucc, Milan, MI
  - Ospedale Civile - Unita' Operativa Di Cardiologia, Rho, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale San Pellegrino - U.O. Cardiologia, Castiglione delle Stiviere, MN
  - Ospedale Policlinico - Uo Cardiologia, Modena, MO
  - Ospedale Civile Di Baggiovara - U.O. Di Cardiologia, Modena, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ftgm - Stabilimento Di Massa - Uoc Cardiologia Diagn. E Interventistica, Massa, MS
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Ospedale Giovanni Paolo Ii - Utic - Cardiologia, Olbia, OT
  - Ospedale Civico - U.O. Cardiologia, Partinico, PA
  - Ospedale Di Camposampiero - U.O.A. Cardiologia, Camposampiero, PD
  - Ospedale Di Cittadella - U.O. Cardiologia, Cittadella, PD
  - Ospedali Riuniti Padova Sud - U.O.C. Cardiologia, Monselice, PD
  - Ospedale Civile Immacolata Concezione - Cardiologia E Utic, Piove di Sacco, PD
  - Ospedale Civile San Massimo - Ambulatorio Di Cardiologia, Penne, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Di Cardiologia, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista - S.C. Cardiologia, Foligno, PG
  - Ospedale Della Val Di Nievole - U. O. Cardiologia - Utic, Pescia, Point
  - Ospedale San Jacopo - U.O. Cardiologia, Pistoia, Point
  - Fondazione Irccs Policlinico San Matteo - Card. Con Ucc-Lab. Ricerca Sperim. Card., Pavia, PV
  - Ospedale Civile - Cardiologia, Vigevano, PV
  - Ospedale S. Giovanni Di Dio - U.O. Cardiologia E Utic, Melfi, PZ
  - Azienda Ospedaliera San Carlo - Uo Cardiologia Utic E Cardiostimolazione, Potenza, PZ
  - Ospedale Civile - S.O.C. Cardiologia-Utic, Locri, RC
  - Ospedale Santa Maria Degli Ungheresi - U.O. Di Cardiologia, Polistena, RC
  - Ao Bianchi Melacrino Morelli- Po Riuniti - Divisione Di Cardiologia, Reggio Calabria, RC
  - Policlinico Madonna Della Consolazione - U.O. Di Cardiologia, Reggio Calabria, RC
  - Ospedale Civile San Sebastiano - Sos Cardiologia Area Nord, Correggio, RE
  - Ospedale Civile - Sc Cardiologia Area Nord, Guastalla, RE
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia, RE
  - Ospedale Riccardo Guzzardi - U.O.C. Di Cardiologia-Utic, Vittoria, RG
  - Aslrm6-Polo H2 Albano-Genzano - U.O.C. Di Cardiologia E Utic, Albano Laziale, RM
  - Ospedale Civile San Paolo - U.O. Cardiologia - Utic, Civitavecchia, RM
  - Ospedale L. Parodi Delfino - U.O. Complessa Di Cardiologia - Utic, Colleferro, RM
  - Ospedale San Sebastiano Martire - U.O. Cardiologia - Utic, Frascati, RM
  - Policlinico Citta' Di Pomezia S. Anna - U.O. Cardiologia-Utic, Pomezia, RM
  - Campus Biomedico - Cardiologia, Roma, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia 1, Roma, RM
  - Policlinico Umberto Primo - Cardiologia B - Cardiologia E Angiologia, Roma, RM
  - Aurelia Hospital - U.O.C Cardiologia, Roma, RM
  - Policlinico Agostino Gemelli - Cardiologia Intensiva, Roma, RM
  - Ao San Giovanni Addolorata - Cardiologia E Riab. Cardiologica, Roma, RM
  - Ospedale Fatebenefratelli - U.O.C. Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Casa Di Cura Madonna Della Salute - Cardiologia, Porto Viro, RO
  - Ospedale Santa Maria Della Misericordia - U.O.C. Cardiologia, Rovigo, RO
  - Presidio Osped. S. Maria Della Speranza - U.O. Di Cardiologia, Battipaglia, SA
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Ospedale G. Fucito - U.O. Di Cardiologia E Utic, Mercato San Severino, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Cardiologia Interventistica - Emodinamic, Salerno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Ospedali Riuniti Della Valdichiana Senese - Cardiologia E Utic, Montepulciano, SI
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Ospedale Civile - U.O. Cardiologia, Sondrio, SO
  - Ospedale San Bartolomeo - U.O. Cardiologia Clinica-Riabilitativa, Sarzana, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - Ospedale Civile M. Giannuzzi - Cardiologia E Utic, Manduria, TA
  - Ospedale Ss. Annunziata - S.C. Cardiologia-Utic, Taranto, TA
  - Ospedale Civile G. Mazzini - Cardiologia Utic Ed Emodinamica, Teramo, TE
  - Ospedale Santa Maria Del Carmine - Cardiologia, Rovereto, TN
  - Por Cirie'- Lanzo Presidio Cirie' - S.C. Cardiologia Cirie'- Ivrea, Cirié, TO
  - Ospedale Civile - S.C. Cardiologia Cirie' Ivrea, Ivrea, TO
  - Ospedale Degli Infermi - Sc Cardiologia, Rivoli, TO
  - Ospedale Ss. Vito E Spirito - U.O.S. Di Cardiologia, Alcamo, TP
  - Ospedale S. Maria Della Stella - Sc Di Cardiologia, Orvieto, TR
  - Azienda Ospedaliera Santa Maria - S.C. Di Cardiologia, Terni, TR
  - Ospedali Riuniti - Osp. Cattinara - S.O.C. Cardiologia, Trieste, TS
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Ospedale S. Antonio Abate - U.O. Di Cardiologia, Gallarate, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo Galmarini - Cardiologia, Tradate, VA
  - Ospedale Di Circolo E Fondazione Macchi - Cardiologia I, Varese, VA
  - Ospedale Di Circolo E Fondazione Macchi - Ssd Unita' Di Cure Intensive Coronariche, Varese, VA
  - Ospedale Dell'Angelo - U.O. Cardiologia, Mestre, VE
  - Ospedale Civile - Ambulatori Cardiologia, Portogruaro, VE
  - Ospedale Civile Di Venezia - U.O. Di Cardiologia, Venezia, VE
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Ospedale San Bassiano - Struttura Complessa Di Cardiologia, Bassano del Grappa, VI
  - Ospedale Alto Vicentino - U.O.C. Cardiologia - Ucic, Santorso, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Giugliano in Campania
  - Ospedale Buon Consiglio Fatebenefratelli - U.O.Complessa Di Cardiologia E Utic, Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi - U.O.C. Cardiologia - S.U.N., Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi - U.O.C. Cardiologia, Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic, Napoli
  - Fondazione Evangelica Betania - Uos Cardiologia, Napoli
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara
  - Casa Di Salute Santa Lucia - U.O. Cardiologia, San Giuseppe Vesuviano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulizia MM, Cemin R, Colivicchi F, De Luca L, Di Lenarda A, Boriani G, Di Pasquale G, Nardi F, Scherillo M, Lucci D, Fabbri G, Maggioni AP; BLITZ-AF Investigators. Management of atrial fibrillation in the emergency room and in the cardiology ward: the BLITZ AF study. Europace. 2019 Feb 1;21(2):230-238. doi: 10.1093/europace/euy166. PMID 30060174
- [Result] Cemin R, Colivicchi F, Maggioni AP, Boriani G, De Luca L, Di Lenarda A, Di Pasquale G, Fabbri G, Lucci D, Gulizia MM; On the behalf of BLITZ-AF Investigators. One-year clinical events and management of patients with atrial fibrillation hospitalized in cardiology centers: Data from the BLITZ-AF study. Eur J Intern Med. 2020 Apr;74:55-60. doi: 10.1016/j.ejim.2019.12.006. Epub 2020 Jan 14. PMID 31952984